CLINICAL TRIAL: NCT00497237
Title: Prospective, Randomised, Open-label, Multicentre, Active Drug Controlled, Parallel Group Design Clinical Trial of the Efficacy and Safety of Beclomethasone Dipropionate 400 mcg + Formoterol 24 mcg pMDI Via HFA-134a (Foster™) vs. Fluticasone Propionate 500 mcg + Salmeterol Xinafoate 100 mcg DPI (Seretide Diskus®) in the 6 Months Stepdown Treatment of Adult Patients With Controlled Asthma
Brief Title: Clinical Trial of the Efficacy and Safety of Beclomethasone Dipropionate Plus Formoterol vs Fluticasone Propionate Plus Salmeterol in the 6 Months Step Down Treatment of Asthma
Acronym: FORTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Gabriele Nicolini, Chiesi Farmaceutici
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC/PR/033011/005/06; 2006-005349-13 (EudraCT Number)
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma; Stepdown; Beclomethasone; Formoterol; Corticosteroids
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Foster
  Interventions: Drug: Beclomethasone plus formoterol fixed combination
- 2 (Active Comparator): Seretide
  Interventions: Drug: Fluticasone plus salmeterol fixed combination

INTERVENTIONS:
Drug: Beclomethasone plus formoterol fixed combination — 100+6 pMDI
  Arms: 1
Drug: Fluticasone plus salmeterol fixed combination — diskus 250/50
  Arms: 2

SUMMARY:
Asthma is a serious global health problem. People of all ages in countries throughout the world are affected by this chronic airway disorder that can be severe and sometimes fatal. The prevalence of asthma is increasing everywhere, especially among children.According to international guidelines, once control of asthma is achieved and maintained for at least 3 months, a gradual reduction of the maintenance therapy should be tried in order to identify the minimum therapy required to maintain control. This will help reduce the risk of side effects and enhance patient adherence to the treatment plan.

Reduction of therapy in patients on combination therapy should begin with a reduction in the dose of inhaled glucocorticosteroid.1 The present study is designed to evaluate if patients with controlled asthma treated with FP 1000 mcg + salmeterol 100 mcg daily can be stepped down. Stepping-down will be attempted with two medications: a new combination of extrafine beclomethasone dipropionate 400 mcg + formoterol 24 mcg daily (test medication, Foster™) and, alternatively, fluticasone propionate 500 mcg + salmeterol 100 mcg daily(reference medication) without losing asthma control.If this hypothesis will be confirmed, the present study will demonstrate that asthma control can be maintained with less than half the dose of inhaled corticosteroid and with less medical costs.

Given the aims of this study, the population to be monitored includes adult patients with moderate persistent asthma, which can be defined controlled according to the current guidelines under standard stabilised treatment. The intended treatment duration is therefore designed to ensure that good control of asthma is firmly achieved before stepping down the treatment (8 weeks run-in period), but also that the condition of the patients are followed long enough (24 weeks comparative treatment period) to ensure that a new stable condition is also obtained and properly monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be enrolled for screening at Visit 1 into the run-in period if they meet all the following criteria:
* Clinical diagnosis of moderate persistent asthma for at least 6 months, according to GINA revised version 2005 guidelines 1 and considering current treatment;
* Forced expiratory volume (FEV1) or peak expiratory flow rate (PEFR) ≥ 80% of the predicted normal value;
* Treated with fluticasone 1000 mcg + salmeterol 100 mcg daily for at least 4 weeks at a stable dose;
* Reporting no nocturnal symptoms or awakenings, no exacerbations, no limitations of activities, symptoms in ≤2 days and use of rescue medication ≤2 days per week, in the last 4 weeks;
* Exhibiting a co-operative attitude and ability to be trained to correctly use the study devices and to complete the diary cards.

At the end of run in period (Week 8+0; Visit 3), patients will be recruited into the treatment period and randomized to treatment if they meet the following criterion:

* Asthma is controlled 1 in each of the last 4 weeks of run-in (no nocturnal symptoms or awakenings; no exacerbations; no limitations of activities; symptoms in ≤2 days; use of rescue medication ≤2 days; morning PEF ≥80% of predicted in every day) confirmed by reviewing the diary cards.

Exclusion Criteria:

* Inability to carry out pulmonary function testing;
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) as defined by the NHLBI/WHO's GOLD guidelines;
* Current smokers or recent (less than one year) ex-smokers with a smoking history of ≥10 pack/years;
* History of near fatal asthma;
* Evidence of symptomatic infection of the airways in the previous 8 weeks;
* Three or more courses of oral corticosteroids or hospitalisation due to asthma during the previous 6 months;
* Patients treated with anticholinergics and antihistamines during the previous 2 weeks, with topical or intranasal corticosteroids and leukotriene antagonists during the previous 4 weeks;
* History or current evidence of heart failure, coronary artery disease, myocardial infarction, severe hypertension, cardiac arrhythmias;
* Diabetes mellitus;
* PTCA or CABG during the previous six months;
* Patients with an abnormal QTc interval value in the ECG test, defined as >450 msec in males or > 470 msec in females;
* Other haemodynamic relevant rhythm disturbances (including atrial flutter or atrial fibrillation with ventricular response, bradycardia (≤55 bpm), evidence of atrial-ventricular (AV) block on ECG of more than 1st degree;
* Clinically significant or unstable concurrent diseases: uncontrolled hyperthyroidism, significant hepatic impairment, poorly controlled pulmonary (tuberculosis, active mycotic infection of the lung), gastrointestinal (e.g. active peptic ulcer), neurological or haematological autoimmune diseases;
* Cancer or any chronic diseases with prognosis <2 years;
* History of alcohol or drug abuse;
* Patients treated with monoamine oxidase inhibitors, tricyclic antidepressants or beta-blockers as regular use;
* Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients;
* Patients who received any investigational new drug within the last 12 weeks;

At the end of run in period (Week 8+0; Visit 3), patients will not be randomized to treatment if they do not completely meet the definition of "controlled asthma". These subjects will be considered screening failures and will not count against the planned number to be recruited.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Morning pre-dose PEF measured daily by patients (mean of the last 2 weeks of treatment period). | mean of the last 2 weeks of treatment period

SECONDARY OUTCOMES:
symptom scores and symptom free days | in the whole study period and every 2-week period
morning and evening pre-dose PEF and FEV1 measured daily by patients; | daily and mean each 2-week period
pulmonary function tests measured at clinics (pre-dose PEF, FVC and FEV1); | at aech clinic visit
change of FEV1 from pre-dose to 5, 15, 30 and 60 minutes post-dose; | randomization visit and end of treatment visit
number, frequency and severity of exacerbations, time to first exacerbation | whole study period
adverse events and adverse drug reactions | retrospectively assessed at each visit
use of relief salbutamol and days without use of relief salbutamol; | daily
proportion of patients with controlled asthma and partly controlled asthma, weeks of controlled asthma and partly controlled asthma; | weekly
pharmaco-economic analysis of medical and non medical costs. | during study period
12 h-overnight urinary cortisol/creatinine | (collected at visit 3, 6 and 9)
vital signs | at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Paggiaro, MD, Principal Investigator — Ospedale Cisanello, Pisa
Locations (18):
- Bulgaria (4):
  - Clinic of Pulmonology, UMHAT "Sveti Georgi", Plovdiv
  - First Department of Pulmonology, Regional Dispensery of Pulmonology and Phtisiatric Diseases with Stationary (RDPPDS), Rousse
  - Clinic of Pulmonology, University Hospital "Lozenetz", Sofia
  - First Internal Clinic, Endocrinology and Pulmonology Department MHAT, Stara Zagora
- Italy (4):
  - U.O.C. S.Anna e S. Sebastiano - Malattie dell'apparato respiratorio, Caserta
  - Ospedale S. Camillo de Lellis - U.O.C. Pneumologia, Chieti
  - Ospedale Cardarelli - Fisiopatologia Respiratoria, Napoli
  - CNR - Dipartimento di Fisiopatologia Respiratoria, Palermo
- Ukraine (10):
  - Department of Hospital Pediatrics Crimean State Medical University. Pulmonology Department of Republican Clinical Children's Hospital, Crimea
  - Pulmonological and Allergological Department of the Kharkov Regional Clinical Hospital, Kharkiv
  - Pulmonological Department #2, Kharkiv
  - Pulmonological Department of the Institute of Therapy, Ukrainian Academy of Medical Sciences, Kharkiv
  - Department of General Practice- Family medicine. Medical Academy of postgraduate education., Kharkiv
  - Department of Diagnostic, Therapy and Clinical Pharmacology of Lung Diseases of the Institute of Phthisiology and Pulmonology Academy of Medical Science of the Ukraine, Kiev
  - Institute of pthysiology and pulmonology Academy of medical science of the Ukraine., Kiev
  - Pulmonology Department of the Institute of Phthisiology and Pulmonology AMS of the Ukraine, Kiev
  - Clinical Hospital 8, Department of pediatrics and clinical laboratories, Kryvyi Rih
  - Department of Hospital Therapy of Lugansk State Medical Institute. Lugansk Regional Clinical Hospital, Luhansk

REFERENCES:
- [Result] Papi A, Nicolini G, Crimi N, Fabbri L, Olivieri D, Rossi A, Paggiaro P. Step-down from high dose fixed combination therapy in asthma patients: a randomized controlled trial. Respir Res. 2012 Jun 25;13(1):54. doi: 10.1186/1465-9921-13-54. PMID 22731754
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2006-005349-13